CLINICAL TRIAL: NCT05980312
Title: Early Range of Motion Versus Plaster Immobilization After Open Reduction Internal Fixation of Elbow Fractures: A Prospective, Randomized Trial
Brief Title: Does Early Elbow Motion Improve Patient Outcomes After Surgically Treated Elbow Fractures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, David Fuller, Orthopaedic Surgeon, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-196
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Elbow Fracture; Range of Motion; Immobilization
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Intervention Model Description: Prospective, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilized (Active Comparator): Patients in the control group will be immobilized for 2 weeks and resume unrestricted motion once the splint is taken off.
  Interventions: Other: Splint Immobilization
- Early Range of Motion (Experimental): Patients in the experimental group will start early motion immediately after surgery.
  Interventions: Other: Early Motion

INTERVENTIONS:
Other: Splint Immobilization — Patients will be randomized to receive a splint following their surgical procedure.
  Arms: Immobilized
Other: Early Motion — Patients will be randomized to receive no splint following their surgical procedure.
  Arms: Early Range of Motion

SUMMARY:
The purpose of this study is to compare the safety and efficacy, defined as improved range of motion and functional outcome scores, of early elbow motion in the early (immediately post-op) and late postoperative periods (2 week post-op).

DETAILED DESCRIPTION:
A prospective randomized clinical trial will be performed. Patients over the age of 18 undergoing operative fixation of an elbow fracture by a Cooper orthopaedic surgeon will be considered for study inclusion. Patients who are under the age of 18, pregnant, admitted to the ICU, have a history of trauma/injury to the joint, or extensive soft tissue injury as determined by the treating orthopaedic surgeon will be excluded from study participation. All surgeons listed as co-investigators on this study have agreed to participate. Surgeons who may want to handle postop care differently despite randomization were not listed as co-investigators on this study. All patients will undergo operative fracture fixation of the elbow, which is standard of care. The decision for operative treatment will be made prior to study participation based on fracture classification and the discretion of the orthopaedic trauma team. There are discrete indications for operative treatment of elbow fractures in the orthopaedic literature. These guidelines are based upon the AO/OTA fracture classifications. Operative indications for elbow fractures include: type 13 humerus fractures including all subtypes, type 2r1 radius fractures including all subtypes, and type 2u1 ulna fractures including all subtypes. After this decision is made, the patient will be considered for study inclusion. There will be two treatment groups. The control group will be immobilized in a splint for 2 weeks and will be allowed to resume unrestricted motion at 2 weeks postop. The experimental group will be allowed to use unrestricted motion immediately after surgery. Both groups will be followed up postoperatively to monitor for pain, range of motion, and elbow function as well as the presence of complications. Once there is adequate pain control and if there are no complications, the patient will be discharged. All patients will be instructed to follow up with their surgeon within 2 weeks. If patients do not follow-up with the surgeon in 2 weeks time, the research team will call the patient to monitor clinical progress. At the time of follow-up, all patients will be recommended to go to physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have undergone operative treatment for an elbow fracture
* Operative indications for elbow fractures include: Type 13 humerus fractures including all subtypes, Type 2r1 radius fractures including all subtypes, Type 2u1 ulna fractures including all subtypes.
* Individuals over the age of 18 years old.

Exclusion Criteria:

* Any patient who had not undergone operative treatment of an elbow fracture will be excluded.
* Patients who were not treated surgically by an orthopaedic surgeon or were treated outside of the study frame will be excluded.
* Individuals under the age of 18.
* Pregnant women.
* Patients admitted to the intensive care unit (ICU).
* Patients with a history of trauma or injury to the affected elbow will be excluded.
* Patients with extensive soft tissue injury of the elbow, which is defined as any injury that requires graft coverage, will be excluded.
* Non-English speaking patients will be excluded.
* Decisional-impaired patients will be excluded (as no substitute consent is requested).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
ASES-E Scores | Preoperative and postoperatively as 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  A standardized elbow evaluation was developed by the Research Committee of the American Shoulder and Elbow Surgeons 1 (ASES). This score allows the evaluation of elbow function independently from the underlying diagnosis.
HSS Elbow Score | Preoperative and postoperatively as 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  The Hospital for Special Surgery (HSS) scoring system 31 consists of eight domains described as pain, function, sagittal range, muscle strength, flexion contracture, extension contracture, pronation, and supination.
Range of Motion | Preoperative and postoperatively as 2 weeks, 6 weeks, 3 months, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No